CLINICAL TRIAL: NCT03410199
Title: Ultrasound Evaluation of Inferior Vena Cava Compression During Elective Cesarean Delivery. Comparison of Tilt Versus No Tilt Positioning.
Brief Title: Ultrasound Evaluation of Inferior Vena Cava Compression During Elective Cesarean Delivery.
Status: Completed | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Valerie Zaphiratos, MD, MSc, FRCPC, Assistant Professor, Ciusss de L'Est de l'Île de Montréal
Other Study IDs: 2018-1196
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aortocaval compression by the gravid uterus during the third trimester contributes to decreased venous return to the heart. Neuraxial anesthesia reinforces this hypotension by causing a vasodilatation and venous pooling of blood in the lower limbs. The current practice is to tilt the parturient 15 degrees on the operating table after neuraxial anesthesia in order to decrease this hypotension. Recent meta-analysis suggests there is no conclusive evidence to support the tilt position. The goal of our study is to compare ultrasound vena cava variation measurements in the supine versus the tilt position in third trimester parturients undergoing elective cesarean delivery.

DETAILED DESCRIPTION:
Cesarean delivery (CD) is one of the most currently practiced surgeries in the world. In 2013, surgical deliveries represented 32.4% of births in the United States and 26.9% in Canada. Maternal hypotension is a frequent adverse event during CD under spinal anesthesia and can be detrimental to the fetus and mother. Many means have been studied to decrease the incidence of hypotension in this context such as crystalloid/colloid pre-loading and co-loading, vasopressors, and positioning.

Aortocaval compression of the inferior vena cava (IVC) by the gravid uterus is a major contributor to this hypotension and many positions on the operating table have been researched to decrease its influence.Current recommendations for term women undergoing cesarean delivery include left lateral 15 degree tilt in order to reduce aortocaval compression which may cause maternal hypotension and fetal compromise. However, a recent meta-analysis did not show conclusive evidence to favour the tilted versus the supine position. This is probably due to a compensatory mechanism involving venoconstriction of the lower limbs, raising venous pressure and causing flow through collateral channels. Supine hypotensive syndrome with clinically significant effects occurs in 8-10% of women at term, possibly due to less compensatory mechanisms.

Respiratory variations of the IVC diameter measured by an ultrasound may determine the best position on the operating table for term parturients during cesarean delivery. Large variations of IVC diameter during expiration and inspiration have been shown to be related to hypotension in non-pregnant patients.

The primary objective of our project is to compare the collapsibility index of the inferior vena cava during elective cesarean delivery after the administration of spinal anesthesia with a phenylephrine infusion. Each participant will be their own control.

20 patients scheduled for elective cesarean delivery will be included. Each participant will be her own control for the ultrasound measurements of the inferior vena cava, with and without a tilt before and after spinal anesthesia with a phenylephrine infusion. A transcutaneous oximetry monitor (NIRS) will be used in order to measure the upper versus lower body saturation difference. The newborn Apgar score and umbilical cord pH will be noted.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* Elective cesarean delivery
* Spinal anesthesia
* At least 37 weeks of gestational age
* French speaking patients (able to read and sign the consent form)

Exclusion Criteria:

* Inability to obtain adequate ultrasound mesures before or after spinal anesthesia
* Cardiopathy
* Unexpected difficult spinal anesthesia requiring general anesthesia
* Unexpected complications requiring strong hemodynamic support (transfusions, volume challenges, multiple vasopressors, inotropic drugs...) or requiring anti-hypertensive medication (including magnesium)
* Any contraindication or patient's refusal for spinal anesthesia (e.g. coagulopathy)
* Morbid obesity (IMC over 40 at the time of delivery)
* Active labour
* Emergency cesarean delivery
* Fetal abnormality or prematurity (under 37 weeks of gestational age)
* Multiple gestation
* Inability to cooperate due to langage or physical/mental incapacity

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Third trimester parturients with a normal pregnancy and a planned cesarean delivery under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Collapsibility index of the inferior vena cava after spinal anesthesia. | Day 0
  Comparison of the collapsibility index of the inferior vena cava with and without a tilt after spinal anesthesia.

SECONDARY OUTCOMES:
Collapsibility index of the inferior vena cava before spinal anesthesia. | Day 0
  Comparison of the collapsibility index of the inferior vena cava with and without a tilt before spinal anesthesia.
Calf versus arm transcutaneous saturation | Day 0
  Comparison of the calf versus arm transcutaneous saturation values in the tilt versus supine positions before and after spinal anesthesia
Impact of the tilt versus no tilt positioning on the Apgar score | 1 hour
  Comparison of the Apgar scores of the newborn in regards to the mother's position on the operating table during the C-section: tilt versus supine.
Impact of the tilt versus no tilt positioning on the umbilical cord pH | 1 month
  Comparison of the umbilical cord pH of the newborn in regards to the mother's position on the operating table during the C-section: tilt versus supine.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Zaphiratos, MD, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Maisonneuve-rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gagne MP, Richebe P, Loubert C, Drolet P, Gobert Q, Denault A, Zaphiratos V. Ultrasound evaluation of inferior vena cava compression in tilted and supine term parturients. Can J Anaesth. 2021 Oct;68(10):1507-1513. doi: 10.1007/s12630-021-02051-w. Epub 2021 Jul 1. PMID 34212308